CLINICAL TRIAL: NCT06639399
Title: Effect of Acupuncture at Different Combinations of Acupoints for Postoperative Urinary Retention After Radical Hysterectomy of Cervical Cancer: a Retrospective Cohort Study
Brief Title: Effect of Different Acupuncture Schemes for Postoperative Urinary Retention in Cervical Cancer Patients
Status: Completed | Type: Observational
Sponsor: Lu Chao (Other)
Responsible Party: Sponsor-Investigator, Lu Chao, Clinical Professor, Zhejiang Cancer Hospital
Organization: Zhejiang Cancer Hospital (Other)
Other Study IDs: IIT-2024-385
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Urinary Retention (POUR)
MeSH Terms: interventions — Acupuncture Therapy; Electroacupuncture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Patients received acupuncture treatment at the lumbosacral region, all acupoints belong to the bladder meridian, including Shenshu (BL23), Pangguangshu (BL28), Ciliao (BL32), Huiyang (BL35), and Zhibian (BL54) selected bilaterally.
  Interventions: Other: Acupuncture
- Group B: Patients received acupuncture treatment using a comprehensive acupoint combination scheme. In addition to the acupoints used in Group A, the following acupoints were added: Qihai (RN6), Guanyuan (RN4), Zhongji (RN3), Shuidao (ST28), Yinglingquan (S9), and Sanyinjiao (SP6).
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Patients received acupuncture treatment at the lumbosacral region, all acupoints belong to the bladder meridian, including Shenshu (BL23), Pangguangshu (BL28), Ciliao (BL32), Huiyang (BL35), and Zhibian (BL54) selected bilaterally. Electroacupuncture (EA) was applied to the BL32 and BL54 acupoints at a frequency of 2/100Hz. Each treatment lasting for 30 minutes. Patients received five acupuncture treatments per week for two consecutive weeks
  Other Names: Electroacupuncture
  Groups: Group A
Other: Acupuncture — Patients received acupuncture treatment using a comprehensive acupoint combination scheme. In addition to the acupoints used in Group A, the following acupoints were added: Qihai (RN6), Guanyuan (RN4), Zhongji (RN3), Shuidao (ST28), Yinglingquan (S9), and Sanyinjiao (SP6). The acupuncture and EA procedure for the lumbosacral acupoints was the same as in Group A. After 30 minutes of treatment, abdominal and lower limb acupoints were selected for an additional 30 minutes treatment.Each treatment lasting for 60 minutes.Patients received five acupuncture treatments per week for two consecutive weeks
  Other Names: Electroacupuncture
  Groups: Group B

SUMMARY:
This is a retrospective cohort study using a paired control design. We will review the patients of PUR after cervical cancer surgery who went to the acupuncture department and the urinary retention department in Zhejiang Cancer Hospital from October 2020 to August 2024, and 73 patients met the screening criteria. All patients provided written informed consent. The purpose of the study is to compare the effect of acupuncture at different combinations of acupoints for postoperative urinary retention (PUR) after radical hysterectomy of cervical cancer. All outcome-measures data were obtained from past medical records. It is an observational study rather than an intervention study. 73 patients met the screening criteria. They will be assigned into two groups according to the treatment scheme of acupoints combination for acupuncture: Group A (37 cases) and Group B (36 cases).

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* Karnofsky Performance Scale (KPS) score > 70
* met the diagnostic criteria of PUR
* no history of serious urinary system diseases or urinary retention before the operation
* had clear cognition and no severe mental diseases
* had complete medical records and records of residual urine volume data.

Exclusion Criteria:

* presence of other serious systemic diseases or advanced cachexia
* obstructive urinary retention caused by urethral stricture, stones, or other diseases
* receiving other treatments or self-change treatment
* poor compliance or failure to complete the acupuncture treatments
* incomplete clinical data.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of postoperative urinary retention after radical hysterectomy of cervical cancer
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
The change value in residual urine volume | baseline and 2 weeks
  Residual urine volume was assessed before the first treatment and after the final treatment by a trained outpatient nurse using a direct measurement method involving catheter insertion for urine drainage and measurement. Calculate the difference value in residual urine volume before and after treatment.

SECONDARY OUTCOMES:
The patient's abdominal distension sensation by the visual analog scale (VAS) method | baseline and 2 weeks
  Patients were asked to mark their level of abdominal distension sensation on the line, with 0 indicating no abdominal distension and 10 indicating extremely severe abdominal distension.
The occurrence of urinary tract infections | baseline and 2 weeks
  Count the number of urinary tract infections and calculate the incidence rate
The total effective rate | 2 weeks
  Clinical efficacy was assessed based on the change in residual urine volume before and after treatment. Cured: the residual urine volume was significantly decreased and less than 100 ml after treatment, and the catheter was removed with no recurrence during follow-up; Improved: the residual urine volume remained over 100 ml, but decreased by more than 100 ml compared to before treatment; Unimproved: the residual urine volume did not significantly decreased (less than 100 ml) or worsened. The total effective rate was calculated as the number of cured and improved patients divided by the total number of patients×100%.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No